CLINICAL TRIAL: NCT04927975
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study to Evaluate the Safety and Efficacy of Upadacitinib in Subjects With Non-Segmental Vitiligo
Brief Title: Study to Evaluate Adverse Events and Change in Disease Activity With Oral Tablets of Upadacitinib in Adult Participants With Non-Segmental Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-051; 2021-000081-15 (EudraCT Number)
Record Dates: First submitted 2021-06-11; First posted 2021-06-16 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Non-Segmental Vitiligo
Keywords: Vitiligo; Non-segmental vitiligo (NSV); Upadacitinib; ABT-494; RINVOQ
MeSH Terms: conditions — Vitiligo | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Upa 22 mg Period 1, then Upa 22 mg Period 2 (Experimental): Participants received upadacitinib 22 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 22 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2.
  Interventions: Drug: Upadacitinib
- Upa 11 mg Period 1, then Upa 11 mg Period 2 (Experimental): Participants received upadacitinib 11 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 11 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2.
  Interventions: Drug: Upadacitinib
- Upa 6 mg Period 1, then Upa 6 mg Period 2 (Experimental): Participants received upadacitinib 6 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 6 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2.
  Interventions: Drug: Upadacitinib
- Placebo Period 1, then Upa 22 mg Period 2 (Experimental): Participants received Placebo for upadacitinib administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 22 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Placebo Period 1, then Upa 11 mg Period 2 (Experimental): Participants received Placebo for upadacitinib administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 11 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Oral tablets
  Other Names: ABT-494; RINVOQ
Drug: Placebo — Oral tablets
  Arms: Placebo Period 1, then Upa 11 mg Period 2; Placebo Period 1, then Upa 22 mg Period 2

SUMMARY:
Vitiligo is a common chronic autoimmune disease that causes the body's immune system to attack its own pigment producing skin cells. This study is to evaluate how safe and effective upadacitinib is in participants with non-segmental vitiligo. Adverse effects and change in disease activity will be assessed.

Upadacitinib is being evaluated for the treatment of non-segmental vitiligo. The study will enroll approximately 160 participants aged 18-65 with non-segmental vitiligo in 5 treatment arms across 35 sites worldwide.

Participants will either receive study drug vs placebo oral tablets once daily (QD) for 24 weeks (Period A). In Period B (up to 52 weeks), participants who received placebo during the first 24 weeks will switch to study drug. Participants who received study drug during the first 24 weeks, will continue to receive study drug.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-segmental vitiligo (NSV) and no segmental or localized vitiligo.
* Participants with all of the following at Screening and Baseline.

  * Visits: ≥ 0.5 F-VASI and ≥ 5 total vitiligo area scoring index (T-VASI).
  * Participants who have had prior exposure to immunomodulatory biologic therapy, for any indications, but discontinued the biologic therapy prior to the first dose of study drug. Recommended washout periods for biologic therapies include ≥ 4 weeks for etanercept; ≥ 8 weeks for adalimumab, infliximab, certolizumab, golimumab, abatacept, tocilizumab, and ixekizumab; ≥ 16 weeks for secukinumab; and ≥ 12 weeks for ustekinumab. For biologic therapies not specified, therapies must be discontinued at least 5 times the mean terminal elimination half-life of a drug or 3 months prior to Baseline, whichever is longer.

Exclusion Criteria:

* Participants with segmental or localized vitiligo.
* Participants with other skin conditions that would interfere with evaluation of vitiligo, participants with uncontrolled thyroid disease, and participants with > 33% leukotrichia on the face or > 33% leukotrichia on the body (including face).
* Participants previously treated with any topical or systemic janus kinase (JAK) inhibitor or permanent skin bleaching agents.
* Participants treated with any systemic vitiligo therapy (e.g., methotrexate, mycophenolate mofetil, corticosteroids), supplemental vitiligo therapy (antioxidants/vitamins/herbal medicine/traditional Chinese medicine), and/or topical vitiligo therapy including permanent or temporary tattoos within a minimum of 30 days prior to the first dose of study drug (Note: Camouflage and makeup may be used).
* Participants treated with any phototherapy, including excimer (or other forms of laser therapy), within a minimum of 12 weeks prior to the first dose of study drug.
* Participants have history of malignancy other than successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix.
* Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting, and aorto-coronary bypass surgery;
* History of an organ transplant which requires continued immunosuppression;
* History of gastrointestinal (GI) perforation (other than due to appendicitis or mechanical injury), diverticulitis, or significantly increased risk for GI perforation per investigator judgment;
* Conditions that could interfere with drug absorption including but not limited to short bowel syndrome or gastric bypass surgery; subjects with a history of gastric banding/segmentation are not excluded;
* Uncontrolled thyroid disease;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (35):
- United States (20):
  - University of California Irvine /ID# 229390, Irvine, California
  - Stanford University /ID# 228000, Redwood City, California
  - Clearlyderm Dermatology /ID# 227993, Boca Raton, Florida
  - New Horizon Research Center /ID# 229403, Miami, Florida
  - Park Avenue Dermatology, PA /ID# 229400, Orange Park, Florida
  - ForCare Clinical Research /ID# 228010, Tampa, Florida
  - Dawes Fretzin, LLC /ID# 227996, Indianapolis, Indiana
  - Tufts Medical Center /ID# 228087, Boston, Massachusetts
  - Duplicate_UMass Chan Medical School /ID# 228066, Worcester, Massachusetts
  - Duplicate_Michigan Center for Research Company /ID# 228054, Clarkston, Michigan
  - Hamzavi Dermatology /ID# 228056, Fort Gratiot, Michigan
  - Remington-Davis Clinical Research /ID# 229401, Columbus, Ohio
  - Essential Medical Research, LLC /ID# 228074, Tulsa, Oklahoma
  - Oregon Dermatology and Research Center /ID# 228007, Portland, Oregon
  - Oregon Medical Research Center /ID# 228073, Portland, Oregon
  - Duplicate_Medical University of South Carolina /ID# 228067, Charleston, South Carolina
  - International Clinical Research - Tennessee LLC /ID# 228059, Murfreesboro, Tennessee
  - Bellaire Dermatology Associates /ID# 228004, Bellaire, Texas
  - University of Texas Health Science Center at Houston /ID# 229399, Houston, Texas
  - Virginia Clinical Research, Inc. /ID# 228050, Norfolk, Virginia
- Canada (5):
  - Dr. Chih-ho Hong Medical Inc. /ID# 228403, Surrey, British Columbia
  - Wiseman Dermatology Research /ID# 228410, Winnipeg, Manitoba
  - Research Toronto /ID# 228401, Toronto, Ontario
  - Duplicate_K. Papp Clinical Research /ID# 228877, Waterloo, Ontario
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 228388, Québec, Quebec
- France (5):
  - Chu de Nice-Hopital Larchet Ii /Id# 228192, Nice, Alpes-Maritimes
  - Duplicate_Hopital Saint-Andre /ID# 228193, Bordeaux, Gironde
  - HCL - Hopital Edouard Herriot /ID# 228194, Lyon, Rhone
  - Duplicate_Hopital Henri Mondor /ID# 228198, Créteil
  - CHU Toulouse - Hopital Larrey /ID# 228196, Toulouse
- Japan (5):
  - Nagoya City University Hospital /ID# 228725, Nagoya, Aichi-ken
  - Nippon Medical School Hospital /ID# 230361, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 230288, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 230362, Yamagata, Yamagata
  - Yamanashi Prefectural Central Hospital /ID# 229441, Kofu, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Ezzedine K, Soliman AM, Camp HS, Ladd MK, Pokrzywinski R, Coyne KS, Sen R, Schlosser BJ, Bae JM, Hamzavi I. Psychometric Properties and Meaningful Change Thresholds of the Vitiligo Area Scoring Index. JAMA Dermatol. 2025 Jan 1;161(1):39-46. doi: 10.1001/jamadermatol.2024.4534. PMID 39475960
- [Derived] Passeron T, Ezzedine K, Hamzavi I, van Geel N, Schlosser BJ, Wu X, Huang X, Soliman AM, Rosmarin D, Harris JE, Camp HS, Pandya AG. Once-daily upadacitinib versus placebo in adults with extensive non-segmental vitiligo: a phase 2, multicentre, randomised, double-blind, placebo-controlled, dose-ranging study. EClinicalMedicine. 2024 May 31;73:102655. doi: 10.1016/j.eclinm.2024.102655. eCollection 2024 Jul. PMID 38873632
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ITT Population in Period 1 (ITT_1): all randomized participants in Period 1, analyzed according to the treatment groups that they were randomized to. Per protocol, participants who were randomized to Placebo at Baseline were analyzed as one group in Period 1.
  ITT Population in Period 2 (ITT_2): all participants who entered Period 2, analyzed according to the treatment groups that they were randomized to at Baseline.
Groups:
- Placebo Period 1: Participants received Placebo for upadacitinib administered orally once a day (QD) as tablets for 24 weeks during Period 1.
Period: Period 1 (Baseline-Week 24)
Arm/Group | Placebo Period 1 | Placebo Period 1, Then Upa 11 mg Period 2 | Placebo Period 1, Then Upa 22 mg Period 2 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Started | 46 | 0 | 0 | 49 | 47 | 43
Completed | 44 | 0 | 0 | 46 | 45 | 38
Not Completed | 2 | 0 | 0 | 3 | 2 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 2 (Week 24-52)
Arm/Group | Placebo Period 1 | Placebo Period 1, Then Upa 11 mg Period 2 | Placebo Period 1, Then Upa 22 mg Period 2 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Started | 0 | 21 | 22 | 45 | 45 | 33
Completed | 0 | 19 | 21 | 39 | 38 | 30
Not Completed | 0 | 2 | 1 | 6 | 7 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2 | 6 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population in Period 1 (ITT_1): all randomized participants in Period 1, analyzed according to the treatment groups that they were randomized to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2 | Total
Number analyzed (Participants) | 46 | 49 | 47 | 43 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (10.48) | 45.1 (11.68) | 45.5 (11.90) | 48.2 (11.13) | 46.3 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 34 | 26 | 115
  Male | 17 | 23 | 13 | 17 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 4 | 5 | 20
  Not Hispanic or Latino | 41 | 43 | 43 | 38 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 6 | 6 | 7 | 6 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 4 | 3 | 3 | 1 | 11
  White | 34 | 35 | 36 | 33 | 138
  More than one race | 0 | 3 | 1 | 1 | 5
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 4
Total Vitiligo Area Scoring Index (T-VASI) [Mean (Standard Deviation); unit: units on a scale] — The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. It is based on a composite estimate of the overall area of vitiligo patches, measured by the number of hand units (palm plus 5 digits = 1% body surface area [BSA]) multiplied by the degree of depigmentation within each affected area (0%, 10%, 25%, 50%, 75%, 90%, or 100%). The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100, with higher scores indicating more severe disease.
  units on a scale | 21.014 (16.9516) | 20.993 (15.9672) | 22.322 (18.1784) | 21.843 (15.9324) | 21.534 (16.6634)
Facial Vitiligo Area Scoring Index (F-VASI) [Mean (Standard Deviation); unit: units on a scale] — The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3, with higher scores indicating more severe disease.
  units on a scale | 1.043 (0.6094) | 1.154 (0.7655) | 1.021 (0.5781) | 1.159 (0.6585) | 1.094 (0.6559)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Facial-Vitiligo Area Scoring Index (F-VASI) at Week 24
Description: The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3, with higher scores indicating more severe disease. Negative changes from baseline indicate improvement.
Time Frame: Baseline, Week 24
Population: ITT_1: all randomized participants in Period 1, analyzed according to the treatment groups that they were randomized to; mixed model repeated measures analysis (MMRM) including observed measurements at all visits
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Number analyzed (Participants) | 43 | 45 | 43 | 33
Percent change from baseline | -14.36 [-24.86 to -3.85] | -21.96 [-32.18 to -11.75] | -35.63 [-46.11 to -25.14] | -33.96 [-45.41 to -22.50]
Statistical Analysis 1: Comparison: Placebo Period 1 vs Upa 6 mg Period 1, Then Upa 6 mg Period 2; Upa 6 mg Period 1 versus Placebo Period 1; Test type: Superiority — Repeated measures analysis was conducted using a mixed model including observed measurements at all visits. The model included categorical fixed effects of treatment, visit and treatment-by-visit interaction, and stratification factors (age [≤ 50 and > 50], Baseline disease severity [T-VASI < 15 and ≥ 15], active vitiligo [Yes/No]) derived from actual values, and the continuous fixed covariate of Baseline measurement. An unstructured variance covariance matrix was used; p = 0.304, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -7.60, 95% CI 2-sided [-22.18 to 6.97]
Statistical Analysis 2: Comparison: Placebo Period 1 vs Upa 11 mg Period 1, Then Upa 11 mg Period 2; Upa 11 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.005, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -21.27, 95% CI 2-sided [-36.02 to -6.52]
Statistical Analysis 3: Comparison: Placebo Period 1 vs Upa 22 mg Period 1, Then Upa 22 mg Period 2; Upa 22 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.013, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -19.60, 95% CI 2-sided [-35.04 to -4.16]

2. Secondary Outcome: Percentage of Participants Achieving F-VASI 75 (≥ 75% Improvement in F-VASI From Baseline) at Week 24
Description: The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. The F-VASI includes contributions from the face, with a possible range from 0 to 3, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 24
Population: ITT_1: all randomized participants in Period 1, analyzed according to the treatment groups that they were randomized to; NRI-MI (non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 or any other missing data that can be reasonably assumed to be Missing at Random)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Number analyzed (Participants) | 46 | 49 | 47 | 43
percentage of participants | 2.2 [0.0 to 6.4] | 8.2 [0.5 to 15.8] | 19.1 [7.9 to 30.4] | 14.0 [3.6 to 24.3]
Statistical Analysis 1: Comparison: Placebo Period 1 vs Upa 6 mg Period 1, Then Upa 6 mg Period 2; Upa 6 mg Period 1 versus Placebo Period 1; Test type: Superiority — P-value calculated according to the Cochran-Mantel-Haenszel test adjusted for strata (age group [≤ 50 and > 50], baseline disease severity [T-VASI < 15 and ≥ 15], and status of active vitiligo [Yes/No])) for the comparison of two treatment groups. The calculations at each visit were based on non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 or non-responder imputation only if there were no missing data due to COVID-19; p = 0.100, Cochran-Mantel-Haenszel; Response Rate Difference = 6.9, 95% CI 2-sided [-1.3 to 15.2]
Statistical Analysis 2: Comparison: Placebo Period 1 vs Upa 11 mg Period 1, Then Upa 11 mg Period 2; Upa 11 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.002, Cochran-Mantel-Haenszel; Response Rate Difference = 17.8, 95% CI 2-sided [6.5 to 29.0]
Statistical Analysis 3: Comparison: Placebo Period 1 vs Upa 22 mg Period 1, Then Upa 22 mg Period 2; Upa 22 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.026, Cochran-Mantel-Haenszel; Response Rate Difference = 11.7, 95% CI 2-sided [1.4 to 21.9]

3. Secondary Outcome: Percentage of Participants Achieving F-VASI 50 (≥ 50% Improvement in F-VASI From Baseline) at Week 24
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Number analyzed (Participants) | 46 | 49 | 47 | 43
percentage of participants | 10.9 [1.9 to 19.9] | 16.3 [6.0 to 26.7] | 38.3 [24.4 to 52.2] | 39.5 [24.9 to 54.1]
Statistical Analysis 1: Comparison: Placebo Period 1 vs Upa 6 mg Period 1, Then Upa 6 mg Period 2; Upa 6 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.327, Cochran-Mantel-Haenszel; Response Rate Difference = 6.6, 95% CI 2-sided [-6.6 to 19.7]
Statistical Analysis 2: Comparison: Placebo Period 1 vs Upa 11 mg Period 1, Then Upa 11 mg Period 2; Upa 11 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Response Rate Difference = 29.3, 95% CI 2-sided [13.8 to 44.9]
Statistical Analysis 3: Comparison: Placebo Period 1 vs Upa 22 mg Period 1, Then Upa 22 mg Period 2; Upa 22 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Response Rate Difference = 28.7, 95% CI 2-sided [12.6 to 44.7]

4. Secondary Outcome: Percentage of Participants Achieving Total Vitiligo Area Scoring Index (T-VASI) 50 (≥ 50% Improvement in T-VASI From Baseline) at Week 24
Description: The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. It is based on a composite estimate of the overall area of vitiligo patches, measured by the number of hand units (palm plus 5 digits = 1% body surface area [BSA]) multiplied by the degree of depigmentation within each affected area (0%, 10%, 25%, 50%, 75%, 90%, or 100%). The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100, with higher scores indicating more severe disease.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Number analyzed (Participants) | 46 | 49 | 47 | 43
percentage of participants | 2.2 [0.0 to 6.4] | 6.1 [0.0 to 12.8] | 6.4 [0.0 to 13.4] | 11.6 [2.0 to 21.2]
Statistical Analysis 1: Comparison: Placebo Period 1 vs Upa 6 mg Period 1, Then Upa 6 mg Period 2; Upa 6 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.340, Cochran-Mantel-Haenszel; Response Rate Difference = 3.7, 95% CI 2-sided [-3.9 to 11.2]
Statistical Analysis 2: Comparison: Placebo Period 1 vs Upa 11 mg Period 1, Then Upa 11 mg Period 2; Upa 11 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.358, Cochran-Mantel-Haenszel; Response Rate Difference = 3.8, 95% CI 2-sided [-4.3 to 11.8]
Statistical Analysis 3: Comparison: Placebo Period 1 vs Upa 22 mg Period 1, Then Upa 22 mg Period 2; Upa 22 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.027, Cochran-Mantel-Haenszel; Response Rate Difference = 9.1, 95% CI 2-sided [1.0 to 17.2]

5. Secondary Outcome: Percent Change From Baseline in T-VASI at Week 24
Description: The vitiligo area scoring index (VASI) is a validated scoring method used to assess the areas of depigmentation due to vitiligo. It is based on a composite estimate of the overall area of vitiligo patches, measured by the number of hand units (palm plus 5 digits = 1% body surface area [BSA]) multiplied by the degree of depigmentation within each affected area (0%, 10%, 25%, 50%, 75%, 90%, or 100%). The T-VASI is calculated using a formula that includes contributions from all body regions, with a possible range from 0 to 100, with higher scores indicating more severe disease. Negative changes from baseline indicate improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Number analyzed (Participants) | 43 | 45 | 43 | 33
Percent change from baseline | -6.42 [-13.17 to 0.34] | -13.87 [-20.45 to -7.29] | -17.26 [-24.00 to -10.52] | -20.69 [-28.05 to -13.32]
Statistical Analysis 1: Comparison: Placebo Period 1 vs Upa 6 mg Period 1, Then Upa 6 mg Period 2; Upa 6 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.120, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -7.45, 95% CI 2-sided [-16.86 to 1.96]
Statistical Analysis 2: Comparison: Placebo Period 1 vs Upa 11 mg Period 1, Then Upa 11 mg Period 2; Upa 11 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.026, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -10.84, 95% CI 2-sided [-20.37 to -1.32]
Statistical Analysis 3: Comparison: Placebo Period 1 vs Upa 22 mg Period 1, Then Upa 22 mg Period 2; Upa 22 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.005, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -14.27, 95% CI 2-sided [-24.24 to -4.30]

6. Secondary Outcome: Change From Baseline in the Vitiligo Quality-of-Life (VitiQoL) Instrument Total Score at Week 24
Description: The VitiQoL is a validated questionnaire used in clinical trials to assess stigma-related vitiligo impacts. The VitiQoL uses subject-elicited social, affective, and behavior items, asking the subject's appraisal of the vitiligo-related impacts over the last month. Fifteen items are scored on a 7-point scale ranging from 0 ("Not at all") to 6 ("All of the time"). Item scores (0 to 6) are summed to provide a total score range of 0 to 90; higher scores indicate greater impairment of quality of life (QoL). Negative changes from baseline indicate improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
Number analyzed (Participants) | 40 | 44 | 44 | 34
units on a scale | -5.5 [-10.3 to -0.8] | -7.5 [-12.0 to -3.0] | -3.7 [-8.2 to 0.9] | -6.6 [-11.6 to -1.6]
Statistical Analysis 1: Comparison: Placebo Period 1 vs Upa 6 mg Period 1, Then Upa 6 mg Period 2; Upa 6 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.545, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -1.9, 95% CI 2-sided [-8.3 to 4.4]
Statistical Analysis 2: Comparison: Placebo Period 1 vs Upa 11 mg Period 1, Then Upa 11 mg Period 2; Upa 11 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.565, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 1.9, 95% CI 2-sided [-4.5 to 8.3]
Statistical Analysis 3: Comparison: Placebo Period 1 vs Upa 22 mg Period 1, Then Upa 22 mg Period 2; Upa 22 mg Period 1 versus Placebo Period 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.754, Mixed-Effect Model Repeat Measurement; LS Mean Difference = -1.1, 95% CI 2-sided [-7.8 to 5.6]

ADVERSE EVENTS:
Time Frame: All-cause mortality/adverse events were collected from informed consent through the end of the study. Median time on follow-up was 168 days for all groups in Period 1. Median time on follow-up for Period 2 was as follows: Placebo Period 1, Then Upa 11 mg Period 2 (198 days); Placebo Period 1, Then Upa 22 mg Period 2 and Upa 22 mg Period 1, Then Upa 22 mg Period 2 (212 days); Upa 6 mg Period 1, Then Upa 6 mg Period 2 (204 days); and Upa 11 mg Period 1, Then Upa 11 mg Period 2 (207 days).
Groups:
- Placebo Period 1: Participants received Placebo for upadacitinib administered orally once a day (QD) as tablets for 24 weeks during Period 1. AEs and SAEs were collected from the time of informed consent and during Period 1, as long as it did not exceed the start date of Period 2.
- Upa 6 mg Period 1: Participants received upadacitinib 6 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. AEs and SAEs were collected from the time of informed consent and during Period 1, as long as it did not exceed the start date of Period 2.
- Upa 11 mg Period 1: Participants received upadacitinib 11 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. AEs and SAEs were collected from the time of informed consent and during Period 1, as long as it did not exceed the start date of Period 2.
- Upa 22 mg Period 1: Participants received upadacitinib 22 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. AEs and SAEs were collected from the time of informed consent and during Period 1, as long as it did not exceed the start date of Period 2.
- Placebo Period 1, Then Upa 11 mg Period 2: Participants received Placebo for upadacitinib administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 11 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2. AEs and SAEs were collected from the start date of Period 2 to the end of the study.
- Placebo Period 1, Then Upa 22 mg Period 2: Participants received Placebo for upadacitinib administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 22 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2. AEs and SAEs were collected from the start date of Period 2 to the end of the study.
- Upa 6 mg Period 1, Then Upa 6 mg Period 2: Participants received upadacitinib 6 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 6 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2. AEs and SAEs were collected from the start date of Period 2 to the end of the study.
- Upa 11 mg Period 1, Then Upa 11 mg Period 2: Participants received upadacitinib 11 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 11 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2. AEs and SAEs were collected from the start date of Period 2 to the end of the study.
- Upa 22 mg Period 1, Then Upa 22 mg Period 2: Participants received upadacitinib 22 mg administered orally once a day (QD) as tablets for 24 weeks during Period 1. Participants then received upadacitinib 22 mg administered orally once a day (QD) as tablets for 28 weeks during Period 2. AEs and SAEs were collected from the start date of Period 2 to the end of the study.
Arm/Group | Placebo Period 1 | Upa 6 mg Period 1 | Upa 11 mg Period 1 | Upa 22 mg Period 1 | Placebo Period 1, Then Upa 11 mg Period 2 | Placebo Period 1, Then Upa 22 mg Period 2 | Upa 6 mg Period 1, Then Upa 6 mg Period 2 | Upa 11 mg Period 1, Then Upa 11 mg Period 2 | Upa 22 mg Period 1, Then Upa 22 mg Period 2
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/49 | 0/47 | 1/43 | 0/21 | 0/22 | 0/45 | 0/45 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/49 | 0/47 | 3/43 | 1/21 | 0/22 | 0/45 | 2/45 | 0/33
Other Adverse Events (participants affected / at risk) | 26/46 | 19/49 | 28/47 | 23/43 | 9/21 | 11/22 | 12/45 | 22/45 | 17/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Period 1 (N=46) | Upa 6 mg Period 1 (N=49) | Upa 11 mg Period 1 (N=47) | Upa 22 mg Period 1 (N=43) | Placebo Period 1, Then Upa 11 mg Period 2 (N=21) | Placebo Period 1, Then Upa 22 mg Period 2 (N=22) | Upa 6 mg Period 1, Then Upa 6 mg Period 2 (N=45) | Upa 11 mg Period 1, Then Upa 11 mg Period 2 (N=45) | Upa 22 mg Period 1, Then Upa 22 mg Period 2 (N=33)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE LOBULAR BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Period 1 (N=46) | Upa 6 mg Period 1 (N=49) | Upa 11 mg Period 1 (N=47) | Upa 22 mg Period 1 (N=43) | Placebo Period 1, Then Upa 11 mg Period 2 (N=21) | Placebo Period 1, Then Upa 22 mg Period 2 (N=22) | Upa 6 mg Period 1, Then Upa 6 mg Period 2 (N=45) | Upa 11 mg Period 1, Then Upa 11 mg Period 2 (N=45) | Upa 22 mg Period 1, Then Upa 22 mg Period 2 (N=33)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
COVID-19 (Infections and infestations) | 8 (8) | 7 (7) | 9 (9) | 9 (9) | 1 (1) | 5 (5) | 7 (7) | 12 (12) | 5 (5)
GASTROENTERITIS (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 3 (5) | 4 (4) | 2 (2) | 4 (4) | 3 (4) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 4 (4) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 1 (1) | 4 (7) | 2 (3) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
WEIGHT INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 4 (4) | 0 (0) | 9 (11) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 2 (2)
ANXIETY (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 1 (4) | 3 (3) | 4 (4) | 6 (7) | 1 (1) | 2 (3) | 1 (2) | 2 (2) | 3 (3)
DYSHIDROTIC ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT04927975/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT04927975/SAP_001.pdf